CLINICAL TRIAL: NCT00920530
Title: Real-Time PCR for the Detection of Vaginal Group B Streptococcus Carriage at Delivery : a Medico-Economic and Feasibility Study
Brief Title: Real-Time PCR for the Detection of Vaginal Group B Streptococcus Carriage: a Medico-Economic Study
Acronym: BBFAST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, CHU SAINT ETIENNE
Other Study IDs: 0808073
Record Dates: First submitted 2009-06-02; First posted 2009-06-15 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Neonatal Infections; Streptococcus Agalactiae
Keywords: Screening; real time PCR; Streptococcus agalactiae; Pregnant women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Real time PCR monitoring: Women giving birth at the St Etienne Teaching Hospital

SUMMARY:
Group B streptococcus infections may be serious for the neonates. The infection can occur during the birth, by contact with the genital area. That is why the detection of this bacteria is systematically realised in pregnant women between 34 and 37 weeks of amenorrhea in order to give prophylactic antibiotic treatment in case or positive carriage. This strategy presents 2 disadvantages : (1) detection of the group B streptococcus at 34 and 37 weeks of amenorrhea in not predictive of a carriage at delivery, (2) many pregnant women escape from systematic screening, leading to a systematic antibiotic treatment, which means useless costs, and useless antibiotic exposure with resistant bacteria selection. Real time polymerase chain reaction (PCR) allows a rapid detection anytime with no specific microbiological qualification. The aim of the study is to assess the economic outcomes of this strategy and the epidemiological values for St Etienne hospital.

ELIGIBILITY:
Inclusion Criteria:

* women giving birth

Exclusion Criteria:

* planned caesarian
* minor
* cervical diameter > 5 cm
* women giving birth at less than 35 weeks of amenorrhea
* recent antibiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pregnant women having a pregnancy follow up with Streptococcus agalactiae monitoring according with french recommandations.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
number of women receiving a useless antibiotic prevention | 1 day

SECONDARY OUTCOMES:
economic outcomes | 1 day
epidemiological outcomes for group B streptococcus | 1 day
diagnosis efficacy of the real time PCR | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bruno POZZETTO, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France